CLINICAL TRIAL: NCT05659342
Title: Comparison of ELDOA and Mechanical Traction Technique on Pain and Disability in Patients With Lumbar Disc Herniation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Abid ullah
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Lumbar Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ELDOA Technique (Experimental): ELDOA positions (hold for 1 minute, 3 alternative days for 4 weeks). Hot pack (10-15 minutes) McKenzie extension Exercises
  Interventions: Other: ELDOA Technique
- Mechanical Lumbar Traction (Experimental): Mechanical Lumbar Traction (50% of body weight was applied, in supine position, the hip and knee at 90- degree flexion, and the legs were supported.
  Hot pack (10-15 minutes) McKenzie extension Exercises
  Interventions: Other: Mechanical Lumbar Traction

INTERVENTIONS:
Other: ELDOA Technique — the patients treated with ELDOA technique, followed for 3 alternative days for 4 weeks.
  the ELDOA techniques for level L4/L5 and L5/S1 were applied. the ELDOA positions hold for one minute, 3 alternative days for 4 weeks under supervision.
  Hot pack (10-15 minutes) McKenzie Extension Exercises
  Arms: ELDOA Technique
Other: Mechanical Lumbar Traction — Mechanical Traction Technique: traction unit, 50% of body weight was applied with the patients lying in supine position, with the hip and knee at 90 degree flexion, and legs were supported. Traction were applied for 3 alternative days for 4 weeks.
  Hot pack (10-15 minutes) McKenzie Extension Exercises
  Arms: Mechanical Lumbar Traction

SUMMARY:
To compare the effect of ELDOA and Mechanical traction technique on pain in patients with lumbar disc herniation.

To compare the effect of ELDOA and Mechanical traction technique on disability in patients with lumbar disc herniation.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-65 years
* Both gender Male & Female
* Patients having Lumbar radiculopathy diagnosed with lumbar disc herniation.

Exclusion Criteria:

* Patients presented with motor deficit,
* Qauda equina syndrome,
* lumbar fracture
* spinal stenosis,
* osteophyte formation
* facet joint pathology
* spondylolisthesis.
* malignancy,
* degenerative disorders
* recent back surgery and patient whom surgery for lumbar disc herniation/prolapse intervertebral disc already advised by neurosurgeon

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2021-01-04 (Actual); Study Completion 2021-01-04 (Actual)

PRIMARY OUTCOMES:
lumbar ROM by inclinometer. | 4 weeks
  Flexion 60 Extension 25 Left Lat Flex 25 Right Lat Flex 25
pain on Numeric pain rating scale | 4 Weeks
  Changes from baseline, Pain was measured through Numeric pain rating scale.It comprises of a continuous scale of 10cm line.0 to 1 represent no pain, 1 to 3 represent mild pain ,4 to 6 represent moderate pain, 7 to 10 represent severe pain
Modified Oswestry low back pain disability questionnaire | 4th Week
  0% to 20%: minimal disability: The patient can cope with most living activities. Usually no treatment is indicated apart from advice on lifting sitting and exercise. 21%-40%: moderate disability: The patient experiences more pain and difficulty with sitting, lifting and standing. Travel and social life are more difficult and they may be disabled from work. Personal care, sexual activity and sleeping are not grossly affected and the patient can usually be managed by conservative means. 41%-60%: severe disability: Pain remains the main problem in this group but activities of daily living are affected. These patients require a detailed investigation. 61%-80%: crippled: Back pain impinges on all aspects of the patient's life. Positive intervention is required. 81%-100%:These patients are either bed-bound or exaggerating their symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Asghar Khan, DCS-PT, Study Chair — Riphah International University
Locations (1):
- Lady Reading Hospital - Medical Teaching Institution, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No